CLINICAL TRIAL: NCT03062553
Title: Enhancement of Treatment of Delusions in Schizophrenia Through Neuromodulation
Acronym: tACS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Testing for this study remained in the pilot stages due to optimization of the tACS equipment. There are no clinical results to report.
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other); Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Todd Woodward, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H16-01791
Record Dates: First submitted 2016-09-28; First posted 2017-02-23 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Schizophrenia; Psychosis; Delusions
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Delusions | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MCT + Neuromodulation (MCT-N) (Experimental): Participants (n=50) randomly assigned to the MCT-N condition will undergo transcranial alternating current stimulation (tACS) prior to participation in MCT.
  Neuromodulation involving tACS will target increasing the power of the alpha band at dorsomedial prefrontal regions, and this is expected to also decrease the power of the beta band in ventro-medial regions. This will be confirmed by EEG recordings and source estimation during a task.
  The Metacognitive Training (MCT) group intervention will consist of an 8-module cycle occurring twice a week for 4 weeks, for a total of 8 sessions. Each module will include a 45 to 60 minute instructor-led group session using PowerPoint slides and homework assignments to facilitate learning. Groups will consist of 4-10 subjects.
  Interventions: Behavioral: Metacognitive Training (MCT); Device: transcranial alternating current stimulation (tACS)
- Sham/MCT group (MCT- S) (Experimental): Participants (n=50) randomly assigned to the Sham/MCT (MCT-S) condition will undergo the application of random patterns of low-grade currents to the same brain region as the neuromodulation condition prior to participation in MCT.
  MCT is a four week program with eight one-hour sessions. MCT can be obtained online at no cost (www.uke.de/mkt). This experimental intervention will consist of an 8-module cycles occurring twice a week for 4 weeks, for a total of 8 sessions. Each module will include a 45 to 60 minute instructor-led group session using PowerPoint slides and homework assignments to facilitate learning. Groups will consist of 4-10 subjects.
  Interventions: Behavioral: Sham/MCT
- Neuromodulation/Treatment as Usual TAU-N (Experimental): Participants (n=50) randomly assigned to the Neuromodulation/TAU (TAU - N) condition will undergo transcranial alternating current stimulation (tACS) prior to being placed on the TAU waitlist.
  Neuromodulation involving tACS will target increasing the power of the alpha band at dorsomedial prefrontal regions, and this is expected to also decrease the power of the beta band in ventro-medial regions. This will be confirmed by EEG recordings and source estimation during a task.
  TAU is a four week waitlist control group.
  Interventions: Device: transcranial alternating current stimulation (tACS)

INTERVENTIONS:
Behavioral: Metacognitive Training (MCT) — MCT is a group-based program developed directly from current cognitive neuropsychiatry research findings on schizophrenia and psychosis. MCT shares knowledge gained in research labs to help individuals experiencing psychosis become more aware of the thinking patterns involved in their illness. The main purpose of the metacognitive training is to help people change the thinking patterns that cause delusions, thereby avoiding relapse into illness or reducing the impact of delusions.
  Arms: MCT + Neuromodulation (MCT-N)
Behavioral: Sham/MCT — The Sham/MCT group will include application of random patterns of low-grade currents to the same brain region as the neuromodulation condition.
  MCT is a group-based program developed directly from current cognitive neuropsychiatry research findings on schizophrenia and psychosis. MCT shares knowledge gained in research labs to help individuals experiencing psychosis become more aware of the thinking patterns involved in their illness. The main purpose of the metacognitive training is to help people change the thinking patterns that cause delusions, thereby avoiding relapse into illness or reducing the impact of delusions.
  Other Names: Metacognitive Training (MCT)
  Arms: Sham/MCT group (MCT- S)
Device: transcranial alternating current stimulation (tACS) — tACS is a non-invasive brain stimulation technique in which a weak electrical current is applied to the head. The current passing through the brain produces small changes in the excitability of the brain regions falling within the current flow. The current occur in an alternating manner (University of California-Berkeley, 2015).
  Other Names: oscillation-targeted neuromodulation
  Arms: MCT + Neuromodulation (MCT-N); Neuromodulation/Treatment as Usual TAU-N

SUMMARY:
The proposed study aims to use a form of neuromodulation, known as transcranial alternating current stimulation (tACS), to improve the effectiveness of the metacognitive training (MCT) program for treatment of delusions in schizophrenia. tACS is a non-invasive brain stimulation method utilizing weak electrical currents applied to the head to influence neural firing (Antal & Paulus, 2013). Brain regions implicated in delusional thinking will be targeted in the hopes of promoting thinking patterns that will allow participants to question delusional beliefs, reducing the severity of delusions and increasing the positive effects of MCT (Whitman et al., in press; Whitman, Minz & Woodward, 2013). Electroencephalogram (EEG) and behavioural assessments will be used to measure treatment effects.

However, before tACS will be administered to individuals experiencing delusions associated with schizophrenia we will conduct various control-phase (pilot) studies to gain a better understanding on how tACS temporarily alters performance on cognitive processes by biasing dominant patterns of oscillations.

The objective of the pilot studies is to establish the effectiveness of the EGI GTEN system in modulating brain oscillations in the cortex of healthy participants by means of transcranial alternating current stimulation (tACS). In this control/pilot phase of our study, we aim to establish that we can induce changes in the power of a specific frequency band in targeted cortical regions with neuromodulation using the GTEN system, and we will assess whether doing so temporarily alters performance on simple cognitive and perceptual processes in healthy controls. This will be the first step towards translating our stimulation protocol to the patient population for our primary study of interest (tACS as an adjunct to metacognitive training for delusions in psychosis).

DETAILED DESCRIPTION:
Purpose:

The objective of this study is to enhance a form of nonpharmacological treatment of delusions in schizophrenia using neuromodulation, and confirm the effect using electroencephalogram (EEG) and behavioural measures (Whitman et al., in press; Whitman, Minz & Woodward, 2013). Specifically, transcranial alternating current stimulation (tACS) will be used to improve the outcome of participation in metacognitive training (MCT) for the treatment of psychosis.

MCT is a group-based program developed directly from current cognitive neuropsychiatry research findings on schizophrenia and psychosis. MCT shares knowledge gained in research labs to help individuals experiencing psychosis become more aware of the thinking patterns involved in their illness. The main purpose of the metacognitive training is to help people change the thinking patterns that cause delusions, thereby avoiding relapse into illness or reducing the impact of delusions (Moritz et al., 2014).

tACS is a non-invasive brain stimulation technique in which a weak electrical current is applied to the head in order to change the likelihood of neural firing in a region of cortex under the stimulation electrodes (Antal & Paulus, 2013).

Hypothesis:

Neuromodulation will enhance the benefit of the non-pharmacological treatment program, MCT, in the reduction of severity of delusions in schizophrenia.

Justification:

It is now clear that helping individuals with schizophrenia become aware of the thinking patterns that underlie delusions provides effective tools for countering these thinking patterns (Moritz et al., 2013; Mortiz et al., 2014). The MCT program for treatment of delusions involves experiencing situations where everyday interpretations of reality must be questioned. Empirical studies and meta-analyses indicate that MCT is effective, even up to three years after completion of treatment (relative to active control conditions and treatment as usual (TAU)).

Despite these successes, no treatment of schizophrenia can be considered highly effective, and there is always room for improvement in effect size. Neuromodulation can provide this improvement by biasing pathological brain functioning towards a healthy state prior to MCT, enhancing the openness to questioning everyday interpretations of reality, and enhancing the effect of MCT treatment of delusions. tACS is almost entirely non-invasive and purely modulatory, changing the likelihood of neural firing in a region of cortex under the stimulation electrodes. It is now possible to modulate at different frequencies of oscillation, in accordance with how the healthy brain functions when interpreting reality.

The proposed research involves application of oscillation-targeted neuromodulation protocols to bias brain functioning towards a state that promotes questioning everyday interpretations of reality, thereby reducing severity of delusions, and enhancing response to a training program for treatment of delusions in schizophrenia by raising insight about the thinking patterns that lead to delusional thought. The investigators plan to document the brain changes induced by neuromodulation using performance and EEG measures taken on a decision making task that involves interpretation of reality, and for which performance correlates with the severity of delusions. This task involves judging the likelihood that evidence matches a hypothesis, and it has been shown that this judged likelihood increases when patients are strongly delusional. The investigators have shown that this task state (i.e., evidence-hypothesis match) elicits an increase in alpha power in the task positive network, and a decrease in beta power the default-mode network (Whitman et al., in press). This suggests that maximizing the power of the alpha band in the task-positive network should bias the brain towards a healthier state for weighing evidence to test hypotheses about reality, and this can be confirmed with EEG and behavioral measures taken on the aforementioned decision making task, a heightened response to MCT, and a corresponding decrease in the severity of delusions.

Research Design:

Neuromodulation involving tACS will target increasing the power of the alpha band at dorsomedial prefrontal regions, and this is expected to also decrease the power of the beta band in ventro-medial regions. This will be confirmed by EEG recordings and source estimation (Whitman et al., in press; Whitman, Minz & Woodward, 2013). MCT is a four week program with eight one-hour sessions. TAU is a four week waitlist control group. Sham neuromodulation will involve application of random patterns of low-grade currents to the same brain region as the neuromodulation conditions (Antal & Paulus, 2013). Severity of delusions will be measured by the Psychotic Symptom Rating Scales in psychosis (PSYRATS) (Haddock et al., 1999). The behavioral measure of interest is the rating of the match between the evidence and hypothesis, which should decrease as delusions decrease.

Statistical Analysis:

Between-groups (neuromodulation/MCT vs. sham/MCT vs neuromodulation/TAU) analyses of variance (ANOVA) will be carried out on change scores computed on behavioral measures and severity of delusions, pre- and post MCT or TAU, under the hypothesis that decreases in the severity of delusion will be greater in the neuromodulation/MCT condition relative to the sham/MCT and neuromodulation/TAU conditions.

Control-Phase Studies: DREAM Study, Hearing Brain Study and The Effect of Neuromodulation on Saccades Study. Each described below.

Purpose for Control Phase Studies:

The objective of these studies is to establish the effectiveness of the EGI GTEN system in modulating brain oscillations in the cortex of healthy participants by means of transcranial alternating current stimulation (tACS). In this control/pilot phase of our study, we aim to establish that we can induce changes in the power of a specific frequency band in targeted cortical regions with neuromodulation using the GTEN system, and we will assess whether doing so temporarily alters performance on simple cognitive and perceptual processes in healthy controls. This will be the first step towards translating our stimulation protocol to the patient population for our primary study of interest (tACS as an adjunct to metacognitive training for delusions in psychosis).

Justification for Control Phase Studies:

Transcranial alternating current stimulation (tACS) is a non-invasive method used to influence ongoing brain oscillations in humans by applying sinusoidal currents to the scalp (Antal & Paulus, 2013; Vosskuhl, Strüber, & Herrmann, 2018). Human brain oscillations, as measured with electroencephalography (EEG), range from 1 to 100 Hz and are referred to as delta (1-3 Hz), theta (4-8 Hz), alpha (8-12 Hz), beta-1 (13-30 Hz), and gamma (30-40 Hz) oscillations. The oscillations, generated either spontaneously or in response to external stimuli, are the result of rhythmic or repetitive electrical activity of cells, and are known to be involved in the communication of brain regions (Vosskuhl et al., 2018). The synchronization of rhythmical electrical activity leads to increased power in the frequency band of the rhythmical activity. For example, the presentation of an auditory stimulus ("auditory entrainment") at a frequency of 40Hz increases the power of the 40Hz brain oscillations in the auditory cortex ;this phenomenon is known as Auditory Steady-State Response (ASSR; Galambos, Makeig, & Talmachoff, 1981; O'Donnell et al., 2013).

Previous studies have mainly relied on systems that use two large electrodes on the scalp to modulate the underlying brain activity in the oscillation frequency range of interest. The GTEN has 256 potential stimulation sites, as well as advanced source localization techniques, allowing for precise planning and application of current via tailored combinations of electrodes according to the 'reciprocity principle' (Dmochowski, Koessler, Norcia, Bikson, & Parra, 2017; Fernandez-Corazza, Turovets, Luu, Anderson, & Tucker, 2016). The 'reciprocity principal' is a process enabling optimal targeting/stimulation of the brain sources of recorded EEG signal. The GTEN system has in-built software for this very purpose, allowing researchers to program electrodes with the dominant power of frequencies of oscillation, using a small subset of electrodes (4-7) to optimally target the brain regions of interest. This reciprocity principal is ground-breaking in its capacity to demonstrate causal relationships between brain and behavior: by targeting the very brain sources producing brain activity of interest, and applying tACS while observing the behavioral effects on performance (e.g., reaction time, accuracy), one can experimentally link cognitive processes to specific patterns of brain oscillations. Establishing that we are able to use these methods in this way will be an important precursor to our study of tACS as an adjunct to metacognitive training for delusions. Our work using tACS to bias ongoing network activity in the brain rests on being able to accurately target those networks producing the activity of interest, and document whether doing so temporarily changes performance on simple cognitive tasks.

Our "pilot/control" phase with healthy controls will familiarize us with the GTEN system and enable us to optimize the parameters under which GTEN tACS produces short-term changes in cortical excitability and cognitive processes. These insights will inform our larger study focussing on enhancing metacognitive treatment of delusions in schizophrenia using neuromodulation To validate that the GTEN tACS is able to bias ongoing oscillations in targeted cortical areas in a biologically-relevant manner, an initial study in healthy controls ("The Hearing Brain") will investigate the degree to which GTEN tACS applied to the auditory cortex mimics and/or influences the ASSR that endogenously occurs during perception of an auditory tone.

To understand whether GTEN tACS temporarily alters performance on cognitive processes by biasing dominant patterns of oscillations, a second set of initial studies in healthy controls will be run called the "Dynamic Reciprocal Electroencephalography and Modulation (DREAM") study. The DREAM study will apply the reciprocity principle while participants undergo simple cognitive and perceptual tasks. This data collection in healthy controls will include the methods we have already received ethics permission to use with clinical populations (e.g., see 'Enhancement of Treatment of Delusions in Schizophrenia through Neuromodulation Protocol'). Piloting these methods will serve as a verification that tACS can alter cortical excitability in the cortical regions that are implicated in delusional thinking, which we have already been granted permission to neuromodulate in our primary study of patients with schizophrenia. The pilot study will also serve as a preliminary investigation of whether tACS has detectable influences on cognitive tasks that correlate with psychopathology (e.g., delusions). One task involves judging the likelihood that evidence matches a hypothesis, and it has been shown that this judged likelihood increases when patients are strongly delusional.

We also aim to study the behavioural effects of tACS in the "The Effect of Neuromodulation on Saccades Study." Instead of using complex behavioural tasks, we aim to use a simpler and better-understood behaviour response - the oculomotor response. In this study, we aim to use tACS to stimulate the areas involved in oculomotor control to affect eye movements. Participants' gaze will be tracked binocularly using the Eyelink 1,000 system (SR Research, Kanata, ON). The oculomotor response is a well understood behavioural response that is not complex in nature and would allow us to study the effects of tACS on behaviour, this would expand our knowledge on the behavioural effects of tACS. The rationale behind using tACS is that we can target a specific ongoing brain oscillation. In this proof-of-concept study, we plan to use tACS to stimulate frontal eye fields (FEF), which we expect to interrupt the natural network balance, and slow saccades. Thus, the overall objectives of this study are (1) to identify the brain oscillations in FEF underlying saccade preparation and execution, and (2) change activity in these networks through neuromodulation.

Hypothesis:

In the "Hearing Brain" proof-of concept pilot study, we hypothesize that auditory entrainment at 40 Hz as well as GTEN stimulation at 40Hz, but not sham stimulation, will increase the gamma band power in the auditory cortex. Furthermore, we hypothesize stronger gamma band power after GTEN stimulation compared to auditory entrainment.

Regarding the "DREAM studies," we predict that that GTEN applied based on the reciprocity principle will alter participants' accuracy and reaction time while undergoing simple cognitive and perceptual tasks. In particular, regarding the pilot of the methods of the primary study( Enhancement of Treatment of Delusions in Schizophrenia through Neuromodulation), we hypothesize that neuromodulation involving tACS will target increasing the power of the alpha band at dorsomedial prefrontal regions and bias our behavioral measure of interest (the rating of the match between the evidence and hypothesis (see Figure 1 in 'Enhancement of Treatment of Delusions in Schizophrenia through Neuromodulation Protocol').

Regarding the "The Effect of Neuromodulation on Saccades Study," we predict the following: 1. Increased power of alpha oscillation in the FEF will be detected by hdEEG when saccades are execute 2. GTEN-induced alpha oscillations in the FEF will increase saccade latency.

Research Design:

Experimental Design: proof-of concept study "The Hearing Brain"

We will use a between-subjects design to investigate the influence of auditory entrainment, neuromodulation, sham stimulation (control condition), and control frequency stimulation (active control condition) on the power of the gamma band (30-40Hz) in the auditory cortex. All participants will be assigned to either the Neuromodulation, Sham, or Active Control (control frequency) condition, with or without also undergoing the Auditory entrainment condition.

Neuromodulation: For each participant, we will establish a threshold at which the participant first detects the stimulations (e.g., due to phosphenes or skin sensations). In line with other threshold protocols, we will start with tACS stimulation at 40 Hz and 1000 µA for 1 second and increase the amplitude of the stimulation stepwise by 250 µA to a maximum of 3000 µA (Zaehle et al., 2010). Participants will be asked to indicate the presence of any sensations they experience. Each participant's maximum stimulation intensity will be kept 250 µA below their threshold for experiencing phosphenes or skin sensations (whichever threshold is lower).

During stimulation, tACS will be applied over the auditory cortex with a frequency of 40 Hz. For each stimulation, the current will be slowly ramped up to the participant's tailored intensity and ramped down at the end of the segment. The stimulation electrodes in the current proof-of-concept study will be those identified as showing the largest increase in gamma power in an auditory entrainment pilot study.

Auditory entrainment: Participants will be listening to a sequence of tones presented at 40Hz.

Sham: This condition is used to control for expectation effects. Similar to the neuromodulation condition, the current will be ramped up and ramped down; however there will be no stimulation in between.

Control frequency: People in this active control group would be modulated on the same electrodes and with the same current intensity, but at a different frequency band. An active control group is needed in order to make sure the effects are due to the applied frequency of interest and not just due to the current itself.

Rest: After each neuromodulation, entrainment, and sham trial there will be rest period of 50 seconds to measure resting-state EEG.

Each condition ( modulation, sham, auditory entrainment) will be 50 seconds long and presented 7 times in blocks. In between the conditions there will be a 50 seconds resting-state measurement to assess the durability of interventions on brain activity.

Experimental Design: proof-of concept "Dynamic Reciprocal Electroencephalography and Modulation" (DREAM) study

We will use a between-subjects design to investigate the influence of neuromodulation based on the reciprocity principle vs. sham stimulation (control condition) vs. control frequency stimulation (active control condition) on reaction time and accuracy in simple cognitive and perceptual tasks. These tasks include the Stroop Interference Task, listening to/ reading non-offensive non-emotional words, and remembering words or visual arrays.

We also plan to pilot tACS in the evidence-integration task which has been shown to correlate with delusional severity in psychosis. To illustrate the reciprocity principle method for this task, participants will be assigned to receive either tACS or sham neuromodulation. Neuromodulation involving tACS will target the dominant pattern of brain oscillations, which we expect to be the alpha band at dorsomedial prefrontal regions, and doing so is expected to also decrease the power of the beta band in ventro-medial regions (Antal & Paulus, 2013). This will be confirmed by EEG recordings and source estimation (Whitman et al., in press; Whitman, Ward, & Woodward, 2013) during the task used to produce Figure 1. Sham neuromodulation will involve application of random patterns or very brief low-grade currents to the same brain region as the neuromodulation condition (Antal & Paulus, 2013). The behavioral measure of interest in this task is the rating of the match between the evidence and hypothesis (see Figure 1), which has been shown to correlate with delusional severity in psychosis.

Experimental Design: proof-of concept study "The Effect of Neuromodulation on Saccades"

The experiments proposed are standard saccade experiments, similar to the ones conducted by Chen Zhang et al. In the prosaccade task, each trial begins with a fixation point at the center of the screen that lasts for 800-1200 ms picked randomly from an exponential distribution. Participants will be instructed to fixate on the fixation point. The fixation point disappears and, after a time gap of 200 ms, a peripheral target appears randomly at 10° to the left or right of the central fixation point. Participants will be instructed to make a rapid saccade in the direction of the target. They have 1,000 ms to complete the saccade to the correct location. In the anti-saccade task, the procedure remains the same but the participants are instructed to make a saccade in the opposite direction of the target. In the memory-guided saccade task, participants will be instructed to maintain fixation, after which two targets will appear sequentially for 100 ms each in one of four quadrants around the periphery of the screen. Participants will be required to maintain fixation for additional time and wait for the go signal (disappearance of the fixation point). Then the participants are required to make two saccades as accurately as possible to the remembered locations of the targets in the same sequence in which they occurred. The prosaccade, anti-saccade, and memory-guided saccade trials will be interleaved in a block. The different types of tasks will be differentiated by different colors of the fixation cross.

tACS Protocol: All the participants will perform three blocks of the above experiment: pre-stimulation block (pre), stimulation block (stim/sham), post-stimulation block (post). In the pre-stimulation block, participants will perform all the above tasks, simultaneously their EEG data is recorded and their eye-movements are tracked. Based on the EEG data, the exact montage for frontal eye fields (FEF) stimulation will be estimated for each participant. Also, the exact alpha frequency for stimulation will be estimated. Based on these parameters, half the participants will be stimulated in the stimulation block. The other half of the participants will act as controls will undergo a sham block. In both cases, the participants also perform the saccade tasks. The post block is similar to the pre-stimulation block.

Data Analysis:

Proof-of concept study "The Hearing Brain":

Power Spectrum density (PSD) for the range of 1 to 50Hz will be calculated for each of the resting-state measurements and averaged for each of the conditions. Repeated-measures (entrainment vs. neuromodulation vs. sham vs. control frequency) analyses of variance (ANOVA) will be carried out for the PSD values of gamma band and the control frequency bands (alpha, beta), under the hypothesis that neuromodulation and entrainment but not sham will lead to increased gamma band power but not to differences in the control frequencies.

Proof-of-concept "DREAM" study:

Between-groups (neuromodulation vs. sham vs. control frequency stimulation) analyses of variance (ANOVA) will be carried out on change scores computed on behavioral measures (accuracy, reaction time) in order to assess whether tACS applied using the reciprocity principle to bias ongoing brain oscillations alters cognitive performance.

Proof-of concept study "The Effect of Neuromodulation on Saccades":

EEG preprocessing: The hdEEG data recorded using the GTEN system will be analyzed using MATLAB 2019b using in-house scripts. EEGLAB 13.6.5b (Delorme & Makeig, 2004) functions were used to generate the topographical plots. The spectral analysis will be performed using Chronux 2.12 toolbox (Bokil et al., 2010). The EEG data will be preprocessed using a Statistical Correction of Artifacts in Dense-array Studies (SCADS) (Junghöfer et al., 2000), which removes EEG artifacts based on statistical parameters. Firstly, the data will be filtered using an FIR bandpass filter with stop band frequencies at 2Hz and 55Hz. The filter will be designed using the MATLAB based signal processing toolbox. Then the EEG data will be epoched to contain the entire trial. Then, electrodes contaminated with artifacts will be rejected by the SCADS algorithm. The parameters used for electrode rejection are - maximum amplitude, maximum gradient and standard deviation of signal amplitude in each epoch, and each electrode. Further, the EEG data will be re-referenced to the average signal.

Montage estimation using EEG: The exact electrode montage and stimulation frequency to be used in the stimulation block, will be estimated based on the EEG data collected in the pre-stimulation block. The EEG data is preprocessed and epoched w.r.t the saccade onset. EEG data from -1000ms to 500ms from the saccade onset is used to generate epochs. The source of the preparatory activity before the saccade is estimated using Constrained Principal Component Analysis (CPCA) (Takane & Hunter, 2001). CPCA generates a component for the saccade preparation. The electrode loadings for the component will be used as a montage for tACS stimulation. Also, the frequency whose phase encodes the saccade latency (For more details refer to the methods in Drewes & VanRullen, 2011) will be used as the stimulation frequency.

Eye-tracking data analysis: All the data analyses will be performed on MATLAB 2019b. The eye-tracking data will be analyzed using in-house scripts. The eye-tracking data is parsed into different types of epochs. Missing data corresponding to eye-blinks will be rejected from the analysis. Also, the trials in which the participant does not maintain fixation will be rejected. The gaze velocity is used to discriminate saccades from fixations. Then data from each trial is analyzed to check if the participant performed the correct saccade. E.g., if in an anti-saccade trial, the participant saccades away from the target, then the trial is assigned as correct; otherwise, it is assigned as an incorrect trial. Then, for all the trials, behavioral metrics such as saccade accuracy, latency, velocity, amplitude, and trajectories will be extracted. The online effect of stimulation (Stim - Pre) and the long-term effect of stimulation (Post - Pre) is checked for each behavioral metric and each of the saccade tasks. To test hypotheses, analysis of variance (ANOVA) will be carried out on the dependent measures - saccade latency, accuracy, velocity, amplitude, etc, with Sham/Stimulation as the between-subjects variable.

Clinical Impact:

These preliminary studies will be conducted in healthy controls order to establish that we can induce changes in the power of a specific frequency band with neuromodulation using the GTEN system. Further, we aim to establish that we are able to detect short-term changes in EEG signal following tACS and alter cognitive processes that are relevant to the experience of psychiatric illness. Conducting this pilot research will be essential in translating our stimulation protocol to the patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 19 to 60 years with a diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, psychosis not otherwise specified, or a mood disorder with psychotic features will be recruited for this study.

Exclusion Criteria:

* An inability to read and write in English. Participants must be have used English on a daily basis for at least 5 years, and must be able to understand the consent form and give written consent.
* Participants with an IQ score of 80 or lower.
* A history of severe neurological disorder and those with severe manifestations of hostility, megalomania, formal thought disorder and suspiciousness will also be excluded from the analysis.
* Subjects who are consistently disrupting the treatment group might be asked to leave, this will be at the discretion of the group instructor.
* A history of neurological problems (e.g., stroke, aneurysm, Parkinson's, Multiple Sclerosis, encephalitis, meningitis, etc.)
* History of seizure disorder or family history of seizure disorder.
* History of migraines or other types of frequent severe headaches.
* Metallic implants in head.
* Severe head injury, frequent loss of consciousness and/or loss of consciousness greater than 30 minutes.
* Recently suffered a serious concussion
* Pregnancy
* Very fatigued and/or recently experienced severe sleep disturbances
* Medication known to increase risk of stroke and/or seizure.
* Suffer from severe current substance dependence
* Have a psychosis that is a direct consequence of substance abuse

For control-phase studies:

Subjects. We will recruit 440 participants total in the "Enhancement of Treatment of Delusions in Schizophrenia through Neuromodulation" study H16-01791; The current protocol describes the methods to be used in the Control Phase of our research, during which we will recruit 290 healthy controls between 19 and 60 years in order to establish proof-of-concept for using GTEN tACS in modulating brain oscillations and performance on simple cognitive tasks.

Exclusion criteria for healthy controls:

* history of neurological problems (e.g., stroke, aneurysm, Parkinson's, Multiple Sclerosis, encephalitis, meningitis, etc.)
* History of seizure disorder or family history of seizure disorder. While there is no direct evidence to suggest that tACS increases the risk of seizure in those with a history of seizure disorder in their family, research in this area is still relatively recent (< 15 years). Given the unlikely potential for an unknown elevated risk of seizure, we are including this as a conservative precautionary exclusion factor.
* History of migraines or other types of frequent severe headaches. tACS can induce a headache in those prone to migraines and other forms of severe headaches.
* Presence of metallic implants in head.
* History of severe head injury, frequent loss of consciousness and/or loss of consciousness greater than 30 minutes.
* Recent history of a serious concussion
* Current pregnancy.
* Symptoms of severe fatigued and/or recent experience of severe sleep disturbance.
* Medication known to increase risk of stroke and/or seizure

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Psychotic Symptom Rating Scale | 8 weeks post-treatment
  Delusion severity will be measured using the Delusions Scale of the Psychotic Symptom Rating Scales (PSYRATS; Haddock, McCarron, Tarrier, & Faragher, 1999). The PSYRATS Delusion Scale measures specific aspects of delusions such as conviction and impact on thinking.

SECONDARY OUTCOMES:
Scale for the Assessment of Negative Symptoms | 8 weeks post-treatment
  General psychopathology will be assessed using the Scale for the Assessment of Negative Symptoms (SANS; Andreasen, 1984).
Scale for the Assessment of Positive Symptoms | 8 weeks post-treatment
  General psychopathology will be assessed using the Scale for the Assessment of Positive Symptoms (SAPS; Andreasen, 1984).
Signs and Symptoms of Psychotic Illness | 8 weeks post-treatment
  General psychopathology will be assessed using the Signs and Symptoms of Psychotic Illness (SSPI; Liddle et al., 2002).
Jumping to Conclusions Task | 8 weeks post-treatment
  A cognitive biases commonly associated with delusions in schizophrenia will be evaluated using the "jumping to conclusions (JTC) task" (also known as the "fish task"). This task will be carried out on computer tablets. These tasks were developed, in part, by the principal investigator and have been described in previous research (Lecomte & Woodward 2005; Woodward 2006a; Woodward 2006b; Woodward 2007; Moritz & Woodward 2005; Woodward 2009).
Bias Against Disconfirmatory Evidence Task | 8 weeks post-treatment
  A cognitive biases commonly associated with delusions in schizophrenia will be evaluated using the "bias against disconfirmatory evidence (BADE) task". This task will be carried out on computer tablets. These tasks were developed, in part, by the principal investigator and have been described in previous research (Lecomte & Woodward 2005; Woodward 2006a; Woodward 2006b; Woodward 2007; Moritz & Woodward 2005; Woodward 2009).
Electroencephalography Reasoning Bias (Evidence Matching Tasks) | 8 weeks post-treatment
  Subjects will be assessed using electroencephalography (EEG) while they complete tasks in which they must determine whether two pieces of information match, in order to quantify the reactivity of the neural networks believed to be responsible for evidence matching (e.g., anterior-cingulate-based network) and integration of disconfirmatory evidence (bilateral prefrontal-based network). These cognitive bias tasks are the "jumping to conclusions task" (or "fish task") and the "bias against disconfirmatory evidence task" previously described, and were developed in part by the principal investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Todd S Woodward, PhD, Principal Investigator — UBC Professor
Locations (1):
- UBC Hospital - Detwiller Pavilion, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
All data will be reviewed in the aggregate. Individual data will not be analyzed or shared with participants.

REFERENCES:
- [Background] Andreasen NC. The Scale for the Assessment of Negative Symptoms (SANS): conceptual and theoretical foundations. Br J Psychiatry Suppl. 1989 Nov;(7):49-58. No abstract available. PMID 2695141
- [Background] Andreasen NC, Arndt S, Miller D, Flaum M, Nopoulos P. Correlational studies of the Scale for the Assessment of Negative Symptoms and the Scale for the Assessment of Positive Symptoms: an overview and update. Psychopathology. 1995;28(1):7-17. doi: 10.1159/000284894. PMID 7871123
- [Background] Haddock G, McCarron J, Tarrier N, Faragher EB. Scales to measure dimensions of hallucinations and delusions: the psychotic symptom rating scales (PSYRATS). Psychol Med. 1999 Jul;29(4):879-89. doi: 10.1017/s0033291799008661. PMID 10473315
- [Background] Liddle PF, Ngan ET, Duffield G, Kho K, Warren AJ. Signs and Symptoms of Psychotic Illness (SSPI): a rating scale. Br J Psychiatry. 2002 Jan;180:45-50. doi: 10.1192/bjp.180.1.45. PMID 11772851
- [Background] Moritz S, Woodward TS. Jumping to conclusions in delusional and non-delusional schizophrenic patients. Br J Clin Psychol. 2005 Jun;44(Pt 2):193-207. doi: 10.1348/014466505X35678. PMID 16004654
- [Background] Moritz S, Woodward TS. Metacognitive training in schizophrenia: from basic research to knowledge translation and intervention. Curr Opin Psychiatry. 2007 Nov;20(6):619-25. doi: 10.1097/YCO.0b013e3282f0b8ed. PMID 17921766
- [Background] Moritz S, Veckenstedt R, Randjbar S, Vitzthum F, Woodward TS. Antipsychotic treatment beyond antipsychotics: metacognitive intervention for schizophrenia patients improves delusional symptoms. Psychol Med. 2011 Sep;41(9):1823-32. doi: 10.1017/S0033291710002618. Epub 2011 Jan 28. PMID 21275083
- [Background] Woodward TS, Munz M, LeClerc C, Lecomte T. Change in delusions is associated with change in "jumping to conclusions". Psychiatry Res. 2009 Dec 30;170(2-3):124-7. doi: 10.1016/j.psychres.2008.10.020. Epub 2009 Nov 10. PMID 19906443
- [Background] Moritz, S., Veckenstedt, R., Vitzthuma, F., Köthera, U., & Woodward,T.S., Metacognitive training in schizophrenia. Theoretical rationale and administration, in Social Cognition In Schizophrenia: From Evidence to Treatment, David L. Roberts and D.L. Penn, Editors. 2013, Oxford University Press: Oxford. p. 358-383.
- [Background] Moritz S, Veckenstedt R, Andreou C, Bohn F, Hottenrott B, Leighton L, Kother U, Woodward TS, Treszl A, Menon M, Schneider BC, Pfueller U, Roesch-Ely D. Sustained and "sleeper" effects of group metacognitive training for schizophrenia: a randomized clinical trial. JAMA Psychiatry. 2014 Oct;71(10):1103-11. doi: 10.1001/jamapsychiatry.2014.1038. PMID 25103718
- [Background] Whitman JC, Takane Y, Cheung TPL, Moiseev A, Ribary U, Ward LM, Woodward TS. Acceptance of evidence-supported hypotheses generates a stronger signal from an underlying functionally-connected network. Neuroimage. 2016 Feb 15;127:215-226. doi: 10.1016/j.neuroimage.2015.12.011. Epub 2015 Dec 15. PMID 26702776
- [Background] Whitman JC, Ward LM, Woodward TS. Patterns of Cortical Oscillations Organize Neural Activity into Whole-Brain Functional Networks Evident in the fMRI BOLD Signal. Front Hum Neurosci. 2013 Mar 14;7:80. doi: 10.3389/fnhum.2013.00080. eCollection 2013. PMID 23504590
- [Background] Speechley WJ, Whitman JC, Woodward TS. The contribution of hypersalience to the "jumping to conclusions" bias associated with delusions in schizophrenia. J Psychiatry Neurosci. 2010 Jan;35(1):7-17. doi: 10.1503/jpn.090025. PMID 20040242
- [Background] Sanford N, Lecomte T, Leclerc C, Wykes T, Woodward TS. Change in jumping to conclusions linked to change in delusions in early psychosis. Schizophr Res. 2013 Jun;147(1):207-208. doi: 10.1016/j.schres.2013.02.042. Epub 2013 Apr 3. No abstract available. PMID 23561297
- [Background] Cohen J. A power primer. Psychol Bull. 1992 Jul;112(1):155-9. doi: 10.1037//0033-2909.112.1.155. PMID 19565683
- [Background] Antal A, Paulus W. Transcranial alternating current stimulation (tACS). Front Hum Neurosci. 2013 Jun 28;7:317. doi: 10.3389/fnhum.2013.00317. Print 2013. PMID 23825454
- [Background] Woodward TS, Jung K, Hwang H, Yin J, Taylor L, Menon M, Peters E, Kuipers E, Waters F, Lecomte T, Sommer IE, Daalman K, van Lutterveld R, Hubl D, Kindler J, Homan P, Badcock JC, Chhabra S, Cella M, Keedy S, Allen P, Mechelli A, Preti A, Siddi S, Erickson D. Symptom dimensions of the psychotic symptom rating scales in psychosis: a multisite study. Schizophr Bull. 2014 Jul;40 Suppl 4(Suppl 4):S265-74. doi: 10.1093/schbul/sbu014. PMID 24936086
- [Background] Rjosk V, Kaminski E, Hoff M, Gundlach C, Villringer A, Sehm B, Ragert P. Transcranial Alternating Current Stimulation at Beta Frequency: Lack of Immediate Effects on Excitation and Interhemispheric Inhibition of the Human Motor Cortex. Front Hum Neurosci. 2016 Nov 3;10:560. doi: 10.3389/fnhum.2016.00560. eCollection 2016. PMID 27857687
- [Background] Bokil H, Andrews P, Kulkarni JE, Mehta S, Mitra PP. Chronux: a platform for analyzing neural signals. J Neurosci Methods. 2010 Sep 30;192(1):146-51. doi: 10.1016/j.jneumeth.2010.06.020. Epub 2010 Jul 15. PMID 20637804
- [Background] Delorme A, Makeig S. EEGLAB: an open source toolbox for analysis of single-trial EEG dynamics including independent component analysis. J Neurosci Methods. 2004 Mar 15;134(1):9-21. doi: 10.1016/j.jneumeth.2003.10.009. PMID 15102499
- [Background] Dmochowski JP, Koessler L, Norcia AM, Bikson M, Parra LC. Optimal use of EEG recordings to target active brain areas with transcranial electrical stimulation. Neuroimage. 2017 Aug 15;157:69-80. doi: 10.1016/j.neuroimage.2017.05.059. Epub 2017 May 31. PMID 28578130
- [Background] Drewes J, VanRullen R. This is the rhythm of your eyes: the phase of ongoing electroencephalogram oscillations modulates saccadic reaction time. J Neurosci. 2011 Mar 23;31(12):4698-708. doi: 10.1523/JNEUROSCI.4795-10.2011. PMID 21430168
- [Background] Fernandez-Corazza M, Turovets S, Luu P, Anderson E, Tucker D. Transcranial Electrical Neuromodulation Based on the Reciprocity Principle. Front Psychiatry. 2016 May 27;7:87. doi: 10.3389/fpsyt.2016.00087. eCollection 2016. PMID 27303311
- [Background] Galambos R, Makeig S, Talmachoff PJ. A 40-Hz auditory potential recorded from the human scalp. Proc Natl Acad Sci U S A. 1981 Apr;78(4):2643-7. doi: 10.1073/pnas.78.4.2643. PMID 6941317
- [Background] Junghofer M, Elbert T, Tucker DM, Rockstroh B. Statistical control of artifacts in dense array EEG/MEG studies. Psychophysiology. 2000 Jul;37(4):523-32. PMID 10934911
- [Background] Kasten FH, Herrmann CS. Transcranial Alternating Current Stimulation (tACS) Enhances Mental Rotation Performance during and after Stimulation. Front Hum Neurosci. 2017 Jan 31;11:2. doi: 10.3389/fnhum.2017.00002. eCollection 2017. PMID 28197084
- [Background] Parker DA, Hamm JP, McDowell JE, Keedy SK, Gershon ES, Ivleva EI, Pearlson GD, Keshavan MS, Tamminga CA, Sweeney JA, Clementz BA. Auditory steady-state EEG response across the schizo-bipolar spectrum. Schizophr Res. 2019 Jul;209:218-226. doi: 10.1016/j.schres.2019.04.014. Epub 2019 May 9. PMID 31080153
- [Background] Ozen S, Sirota A, Belluscio MA, Anastassiou CA, Stark E, Koch C, Buzsaki G. Transcranial electric stimulation entrains cortical neuronal populations in rats. J Neurosci. 2010 Aug 25;30(34):11476-85. doi: 10.1523/JNEUROSCI.5252-09.2010. PMID 20739569
- [Background] Vosskuhl J, Struber D, Herrmann CS. Non-invasive Brain Stimulation: A Paradigm Shift in Understanding Brain Oscillations. Front Hum Neurosci. 2018 May 25;12:211. doi: 10.3389/fnhum.2018.00211. eCollection 2018. PMID 29887799
- [Background] Zaehle T, Rach S, Herrmann CS. Transcranial alternating current stimulation enhances individual alpha activity in human EEG. PLoS One. 2010 Nov 1;5(11):e13766. doi: 10.1371/journal.pone.0013766. PMID 21072168
- [Background] Zhang C, Paolozza A, Tseng PH, Reynolds JN, Munoz DP, Itti L. Detection of Children/Youth With Fetal Alcohol Spectrum Disorder Through Eye Movement, Psychometric, and Neuroimaging Data. Front Neurol. 2019 Feb 18;10:80. doi: 10.3389/fneur.2019.00080. eCollection 2019. PMID 30833926
- See also: University of California - Berkeley - Committee for Protection of Human Subjects — http://cphs.berkeley.edu/brain_stimulation.pdf
- See also: MCT for Psychosis — http://www.uke.de/mkt
- See also: Constrained principal component analysis: a comprehensive theory. — http://takane.brinkster.net/yoshio/p052.pdf